CLINICAL TRIAL: NCT02390258
Title: A Single Centre, Randomised, Double-blind, Placebo-controlled, Fed-fasted, Single and Multiple Ascending Dose Trial of XEN-D0103 in Healthy Subjects
Brief Title: Fed-Fasted, Single and Multiple Ascending Dose Trial of XEN-D0103
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xention Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XEN-D0103-CL-01
Record Dates: First submitted 2015-03-11; First posted 2015-03-17 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — S66913

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- Part 1: Single Ascending Dose - Cohort 1 (Experimental): 8 subjects (6 receiving 10mg XEN-D0103, 2 receiving placebo)
  Interventions: Drug: 10mg XEN-D0103; Drug: Placebo
- Part 1: Single Ascending Dose - Cohort 2 (Experimental): 8 subjects (6 receiving 30mg XEN-D0103, 2 receiving placebo)
  Interventions: Drug: Placebo; Drug: 30mg XEN-D0103
- Part 1: Single Ascending Dose - Cohort 3 (Experimental): 8 subjects (6 receiving 60mg XEN-D0103, 2 receiving placebo)
  Interventions: Drug: Placebo; Drug: 60mg XEN-D0103
- Part 1: Single Ascending Dose - Cohort 4 (Experimental): 8 subjects (6 receiving 120mg XEN-D0103, 2 receiving placebo)
  Interventions: Drug: Placebo; Drug: 120mg XEN-D0103
- Part 1: Single Ascending Dose - Cohort 5 (Experimental): 8 subjects (6 receiving 200mg XEN-D0103, 2 receiving placebo)
  Interventions: Drug: Placebo; Drug: 200mg XEN-D0103
- Part 2: Fed-Fasted (Experimental): 17 subjects receiving 200mg XEN-D0103 with either a high fat meal or following an overnight fast.
  Interventions: Drug: 200mg XEN-D0103
- Part 3: Multiple Ascending Dose - Cohort 1 (Experimental): 10 subjects (8 receiving 30mg XEN-D0103 twice daily, 2 receiving placebo twice daily)
  Interventions: Drug: Placebo; Drug: 30mg XEN-D0103
- Part 3: Multiple Ascending Dose - Cohort 2 (Experimental): 10 subjects (8 receiving 60mg XEN-D0103 twice daily, 2 receiving placebo twice daily)
  Interventions: Drug: Placebo; Drug: 60mg XEN-D0103
- Part 3: Multiple Ascending Dose - Cohort 3 (Experimental): 10 subjects (8 receiving 150mg XEN-D0103 once daily, 2 receiving placebo once daily)
  Interventions: Drug: Placebo; Drug: 150mg XEN-D0103

INTERVENTIONS:
Drug: 10mg XEN-D0103
  Arms: Part 1: Single Ascending Dose - Cohort 1
Drug: Placebo
  Arms: Part 1: Single Ascending Dose - Cohort 1; Part 1: Single Ascending Dose - Cohort 2; Part 1: Single Ascending Dose - Cohort 3; Part 1: Single Ascending Dose - Cohort 4; Part 1: Single Ascending Dose - Cohort 5; Part 3: Multiple Ascending Dose - Cohort 1; Part 3: Multiple Ascending Dose - Cohort 2; Part 3: Multiple Ascending Dose - Cohort 3
Drug: 30mg XEN-D0103
  Arms: Part 1: Single Ascending Dose - Cohort 2; Part 3: Multiple Ascending Dose - Cohort 1
Drug: 60mg XEN-D0103
  Arms: Part 1: Single Ascending Dose - Cohort 3; Part 3: Multiple Ascending Dose - Cohort 2
Drug: 120mg XEN-D0103
  Arms: Part 1: Single Ascending Dose - Cohort 4
Drug: 200mg XEN-D0103
  Arms: Part 1: Single Ascending Dose - Cohort 5; Part 2: Fed-Fasted
Drug: 150mg XEN-D0103
  Arms: Part 3: Multiple Ascending Dose - Cohort 3

SUMMARY:
This study is an evaluation of the safety and tolerability of XEN-D0103 in healthy subjects. Part 1 assesses the safety, tolerability and blood levels of the ascending single doses of XEN-D0103. Blood levels of XEN-D0103 will be assessed when administered with food and also without food in Part 2. The safety, tolerability and blood levels of XEN-D0103 will be assessed following dosing for 10 days in Part 3.

ELIGIBILITY:
Inclusion Criteria:

* For Parts 1 and 3 healthy, male subjects aged 18 to 45 years, inclusive. For Part 2 healthy, male and female subjects aged 45 to 65 years, inclusive.
* Females must be of non-childbearing potential

Exclusion Criteria:

* Subject has a known heart disease.
* Subject has any of QTcF > 450 msec, PR ≥ 210 msec or QRS ≥ 120 msec at screening (determined from median of three readings).
* For Part 1 only: subject has resting heart rate outside of the range 45 to 80 beats per minute (bpm) at screening (determined from median of three readings).
* Subject has any other condition which, in the investigator's opinion will interfere with the trial.
* Subject has a systolic blood pressure (BP) <80 or >160 mmHg at screening or a diastolic BP >90 or <45 mmHg at screening.
* Subject has a clinically significant abnormal laboratory test result at screening.
* Female subject who is pregnant or breast feeding and female subjects of childbearing potential.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2011-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | Part 1: 13 days; Part 2: 13 days; Part 3: 22 days

SECONDARY OUTCOMES:
Area Under Curve (AUC) of XEN-D0103 following single and multiple dose administration | Part 1: 13 days; Part 3: 22 days
Food effect on AUC of XEN-D0103 | 13 days
Change in QTcF with XEN-D0103 and with placebo | 2 days

CONTACTS AND LOCATIONS:
Locations (1):
- ICON Development Solutions, Manchester, United Kingdom